CLINICAL TRIAL: NCT02665897
Title: Correlation Between Complications of Pre-eclampsia and Detection of Novel Biochemical Markers
Brief Title: Pre-eclampsia and Biochemical Markers
Acronym: PET
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Lecturer, Assiut University
Other Study IDs: PET
Record Dates: First submitted 2016-01-22; First posted 2016-01-28 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Detection of Preeclampsia Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Eclampsia: pregnant women with eclampsia will be diagnosed by the occurrence of seizures on top of preeclampsia.
- severe preeclampsia: pregnant women with severe preeclampsia will be diagnosed according to blood pressure ≥160/110 mmHg with proteinuria detection by boiling method +3,+4.
- healthy: matched normotensive pregnant women.

SUMMARY:
In view of both endothelial injury in pre-eclampsia, high blood pressure and kidney impairment characteristics, a recent study demonstrated that the serum levels of NGAL increased at the end of the second trimester in women who subsequently developed pre-eclampsia compared to the control group.

This correlates well with the endothelial damage that occurs during pre-eclampsia and thus NGAL can be considered as a promising marker in predicting both early and late onset pre-eclampsia. It may be required to combine one or more biomarker with NGAL to increase the precision, and sensitivity for detection of risk and reliability of using biomarkers for pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years.
* Gestational age >20 weeks.

Exclusion Criteria:

* Patients with preexisting renal disease,hypertension, diabetes mellitus, gestational hypertension.
* Patients Refuse to participate in the study
* Patients already have complicated preeclampsia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women after 20 weeks
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The level of circulating NGAL | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes